CLINICAL TRIAL: NCT04916548
Title: Repeated Neurocognitive Measurements in Depressed Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rebecca Price (Other)
Responsible Party: Sponsor-Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21040075
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Ketamine (Experimental): Open-label ketamine infusion
  Interventions: Drug: Intravenous Ketamine

INTERVENTIONS:
Drug: Intravenous Ketamine — Single infusion of intravenous racemic ketamine (0.5mg/kg over 40min)

SUMMARY:
In this project, we will A) track the functioning of a collection of potential neurobiological targets for depression over time, B) examine how fluctuations in the functioning of those targets relates to real-world functioning, and C) in a subset of the sample, determine how the functioning in those targets is altered by a single dose of ketamine.

ELIGIBILITY:
Inclusion Criteria:

All participants will:

1. be between the ages of 18 and 60 years,
2. score ≥ 14 on the Hamilton Depression Rating Scale (Ham-D)
3. possess a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document

Exclusion Criteria:

All participants:

1. Presence of lifetime bipolar, psychotic, or autism spectrum; current problematic substance use (e.g., ongoing moderate-to-severe substance use disorder);
2. Failure to meet standard MRI inclusion criteria: those who have cardiac pacemakers, neural pacemakers, cochlear implants, metal braces, or other non-MRI-compatible metal objects in their body. History of significant injury or surgery to the brain or spinal cord that would impair interpretation of results.
3. Acute suicidality or other psychiatric crises requiring treatment escalation. We will use the Columbia Suicide Severity Rating Scale (CSSRS) as both an initial exclusion criteria (CSSRS "Baseline/Screening" Version for past 1month period) and as grounds for rescue/removal (CSSRS "Since Last Visit" form). The CSSRS will be administered using a paper form by an experienced and thoroughly trained clinical assessor on the study team. Subjects with CSSRS suicide ideation scores scored "yes" on items 4 (active suicidal ideation with some intent to act) and/or 5 (active suicidal ideation with specific plan and intent) will be excluded from the study, and if enrolled, will be exited from the study and referred immediately to the nearest emergency mental health facility for additional thorough assessment and appropriate treatment referral.
4. Changes made to treatment regimen within 4 weeks of baseline assessment.
5. Reading level <6th grade as per patient self-report.
6. Patients who have received ECT in the past 2 months prior to Screening.

Ketamine phase subsample additional exclusion criteria:

1. Patients currently taking any psychotropic medication.
2. Lifetime recreational ketamine or PCP use
3. Current pregnancy or breastfeeding
4. For ketamine phase entry, patients must be reasonable medical candidates for ketamine infusion, as determined by a physician co-investigator. Serious, unstable medical illnesses including respiratory [obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics], cardiovascular [including ischemic heart disease and uncontrolled hypertension], and neurologic [including history of severe head injury] will be exclusions.
5. Clinically significant abnormal findings of laboratory parameters [including urine toxicology screen for drugs of abuse], physical examination, or ECG.
6. Uncontrolled or poorly controlled hypertension, as determined by a physician co-investigator's review of vitals collected during screening and any other relevant medical history/records.
7. Patients with one or more seizures without a clear and resolved etiology.
8. Patients starting hormonal treatment (e.g., estrogen) in the 3 months prior to Screening.
9. Past intolerance or hypersensitivity to ketamine.
10. Patients taking medications with known activity at the NMDA or AMPA glutamate receptor [e.g., riluzole, amantadine, lamotrigine, memantine, topiramate, dextromethorphan, Dcycloserine], or the mu-opioid receptor.
11. Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Ketamine
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.47 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Montgomery-Asberg Depression Rating Scale [Mean (Standard Deviation); unit: score on a scale] — Clinician-rated depression (range: 0-60; higher scores = worse outcome)
  score on a scale | 30.20 (9.29)

OUTCOME MEASURES:

1. Primary Outcome: fMRI Intrinsic Connectivity: Default Mode Network
Description: functional connectivity normalized correlation values within default mode network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.40 (0.11)

2. Primary Outcome: fMRI Intrinsic Connectivity: Frontoparietal Control Network
Description: functional connectivity normalized correlation values within frontoparietal control network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.47 (0.14)

3. Primary Outcome: fMRI Intrinsic Connectivity: Limbic Network
Description: functional connectivity normalized correlation values within limbic network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.44 (0.10)

4. Primary Outcome: fMRI Intrinsic Connectivity: Salience Network
Description: functional connectivity normalized correlation values within salience ventral attentional network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.53 (0.13)

5. Secondary Outcome: fMRI Intrinsic Connectivity: Dorsal Attention Network
Description: functional connectivity normalized correlation values within dorsal attention network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.54 (0.11)

6. Secondary Outcome: fMRI Intrinsic Connectivity: Somatosensory Motor Network
Description: functional connectivity normalized correlation values within somatosensory motor network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.69 (0.10)

7. Secondary Outcome: fMRI Intrinsic Connectivity: Visual Network
Description: functional connectivity normalized correlation values within visual network (range: -1 to +1; larger value = stronger connectivity, smaller value = weaker connectivity)
Time Frame: 24hrs post-intervention
Population: All participants who received a ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
units on a scale | 0.60 (0.08)

8. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
score on a scale | 11.80 (7.55)

9. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
score on a scale | 15.00 (10.45)

10. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 14
score on a scale | 19.93 (13.57)

11. Secondary Outcome: Hamilton Depression Rating Scale (Modified Score)
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
score on a scale | 7.53 (3.89)

12. Secondary Outcome: Hamilton Depression Rating Scale (Modified Score)
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
score on a scale | 11.07 (7.07)

13. Secondary Outcome: Hamilton Depression Rating Scale (Modified Score)
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 14
score on a scale | 13.07 (8.00)

14. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 15
score on a scale | 6.87 (4.60)

15. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 14
score on a scale | 6.79 (4.09)

16. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine
Number analyzed (Participants) | 14
score on a scale | 9.71 (5.59)

17. Other Pre Specified Outcome: Dual Probe Video Task
Description: attentional bias (proportion score) towards sad film clips (range: 0 to +1.0; higher score=greater attention bias towards sad films)
Time Frame: infusion +24 hours (1 day)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Pain Rating Via Quantitative Sensory Testing
Description: Pain rating obtained from Quantitative Sensory Testing by mechanical temporal summation (range: 0-10; higher score=more pain)
Time Frame: 1-hour post-infusion
Reporting Status: Not Posted

19. Other Pre Specified Outcome: PROMIS Pain Intensity Score
Description: PROMIS Pain Intensity Short Form scale T-score (range=0-100; higher score=worse pain)
Time Frame: 1-hour post-infusion
Reporting Status: Not Posted

20. Other Pre Specified Outcome: PROMIS Pain Interference Score
Description: PROMIS Pain Interference Short Form scale T-score (range=0-100; higher score=worse pain)
Time Frame: 1-hour post-infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Adverse events were collected using the Patient Rated Inventory of Side Effects (PRISE; Rush et al 2004) instrument and the Clinician-Administered Dissociative States Scale (CADSS). Open-ended questions were also used to inquire about any additional adverse events not captured on the PRISE. Adverse events were tallied for all symptoms that were reported as new or worsening from pre-infusion baseline with onset during the infusion and/or within the subsequent 24hr period.
Arm/Group | Intravenous Ketamine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Ketamine (N=15)
decreased energy (General disorders) | 1
difficulty sleeping: too little (Psychiatric disorders) | 1
dissociative symptoms (Psychiatric disorders) | 14
dizziness (Nervous system disorders) | 8
dry mouth (Gastrointestinal disorders) | 6
emotional indifference (Psychiatric disorders) | 1
headache (Nervous system disorders) | 1
increased appetite (Gastrointestinal disorders) | 4
loss of sexual desire (Reproductive system and breast disorders) | 1
nausea (Gastrointestinal disorders) | 4
restlessness (General disorders) | 1
sweating (General disorders) | 4
tremors (Nervous system disorders) | 1
trouble achieving orgasm (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT04916548/Prot_SAP_000.pdf